CLINICAL TRIAL: NCT00272701
Title: A Randomised, Open, Phase IV, Parallel Group Multicentre Study to Evaluate a Change of Management in Gastroesophageal Reflux Disease (GERD) Patients by Treatment With Esomeprazole 40 mg or Any Other Proton Pump Inhibitor (PPI), After Initial Treatment Failure, in Ordinary Clinical Practice During 4 Weeks.
Brief Title: Esomeprazole in PPI Failures - IMPROVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00085; IMPROVE; EudraCT-number 2005-000458-57
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2007-08

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole
Drug: Other PPI marketed in Sweden

SUMMARY:
The purpose of this study is to assess how PPI treated GERD patients with insufficient symptom control will benefit from a change in management by providing a more efficient acid secretion inhibition during 4 weeks, by evaluation of esomeprazole 40 mg compared to pre-study PPI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Male or female, aged 18-65 years
* History of GERD symptoms during, at least, six months prior to enrolment
* PPI as maintenance treatment during the last 30 days prior to enrolment
* Heartburn as predominant GERD symptom, as judged by the investigator
* Persisting GERD symptoms during the past 7 days prior to visit 1, judged by the patient as either: 4 days with mild symptoms (i.e. awareness of sign or symptom, but easily tolerated)or 2 days with moderate (i.e. discomfort sufficient to cause interference with normal activities) to severe symptoms (i.e. incapacitating, with inability to perform normal activities)

Exclusion Criteria:

* Any treatment with esomeprazole during 30 days prior to enrolment History of esophageal, gastric or duodenal surgery, except for simple closure of an ulcer
* Current or historical evidence of the following diseases/conditions, as judged by the investigator:Zollinger-Ellison syndrome,Primary esophageal motility disorder, i.e. achalasia, scleroderma, primary esophageal spasm,
* Gastric or duodenal ulcers within the last three months, Malabsorbtion
* Malignancy or other concomitant disease with poor prognosis or which may interfere with the assessments in the study
* Unstable diabetes mellitus. Stable diabetes controlled by diet, oral agents or insulin is acceptable
* Patients with severe diseases or disorders which may interfere with the conduct of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2005-12; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The proportion of patients free from heartburn

SECONDARY OUTCOMES:
Work Productivity and Activity Impairment Questionnaire: Gastro-Esophageal Reflux Disease questionnaire.
EuroQol 5D questionnaire.
Quality Assurance of GERD Treatment Questionnaire
Willingness to pay
Serious Adverse Events and Discontinuations due to Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Sweden Medical Director, MD, Study Director — AstraZeneca
Locations (42):
- Sweden (42):
  - Research Site, Arlöv
  - Research Site, Åkersberga
  - Research site, Bålsta
  - Research Site, Borås
  - Research Site, Bromma
  - Research Site, Bromölla
  - Research Site, Dalby
  - Research Site, Djursholm
  - Research Site, Enskededalen
  - Research Site, Gothenburg
  - Research Site, Grängesberg
  - Research Site, Härnösand
  - Research Site, Helsingborg
  - Research Site, Höllviken
  - Research Site, Jarfalla
  - Research Site, Kil
  - Research Site, Knäred
  - Research Site, Köping
  - Research Site, Kristinehamn
  - Research Site, Linköping
  - Research Site, Ludvika
  - Research Site, Luleå
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Märsta
  - Research Site, Nacka
  - Research Site, Nyköping
  - Research Site, Örebro
  - Research Site, Partille
  - Research Site, Piteå
  - Research Site, Sandviken
  - Research Site, Solna
  - Research Site, Stenstorp
  - Research Site, Stockholm
  - Research Site, Sunne
  - Research Site, Täby
  - Research Site, Trollhättan
  - Research Site, Uppsala
  - Research Site, Varberg
  - Research Site, Varekil
  - Research Site, Vännäs
  - Research Site, Västerås

REFERENCES:
- [Derived] Ekesbo R, Sjostedt S, Sorngard H. Effects of structured follow-up and of more effective acid inhibitory treatment in the management of GORD patients in a Swedish primary-care setting: a randomized, open-label study. Clin Drug Investig. 2011;31(3):181-9. doi: 10.2165/11586330-000000000-00000. PMID 21288053